CLINICAL TRIAL: NCT01144611
Title: A Randomized, Double-blind, Placebo-controlled Phase IIIa Study on bIAP, an Anti-inflammatory Moiety, in Patients Undergoing Combined Aortic Valve Replacement and Coronary Artery Bypass Grafting
Brief Title: Efficacy and Safety of Bovine Intestinal Alkaline Phosphatase (bIAP) During Heart Surgery
Acronym: APPIRED-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alloksys Life Sciences B.V. (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALS-002-2009; 2009-010191-19 (EudraCT Number)
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2011-06

CONDITIONS: Inflammation
Keywords: valve replacement; CABG; SIRTS; Combined aortic valve replacement and CABG surgery
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bIAP (Active Comparator): intravenous as a bolus of bIAP (alkaline phosphatase, 1000 IU) just prior to surgery followed by a 40 IU/kg bIAP infusion during the first 8 hours post surgery.
  Interventions: Drug: bIAP bolus and 8h infusion
- placebo (Placebo Comparator): intravenous as a bolus just prior to surgery followed by an infusion during the first 8 hours post surgery.
  Interventions: Drug: placebo bolus and 8h infusion

INTERVENTIONS:
Drug: bIAP bolus and 8h infusion — intravenous as a bolus of bIAP (bovine intestinal alkaline phosphatase, 1000 IU) just prior to surgery followed by a 40 IU/kg bIAP infusion during the first 8 hours post surgery.
  Arms: bIAP
Drug: placebo bolus and 8h infusion — intravenous as a bolus just prior to surgery followed by an infusion during the first 8 hours post surgery.
  Arms: placebo

SUMMARY:
This multi-centre prospective, randomised, double-blind, placebo-controlled study is designed to evaluate the efficacy and safety of bovine intestinal alkaline phosphatase (bIAP) in reducing the pro-inflammatory post-surgical responses and thereby preserving organ functions in patients undergoing invasive cardiac surgery: combined aortic valve replacement and coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients of any race in the ages of >18 years.
* Patients scheduled for combined aortic valve replacement and CABG surgery.
* Patients who have given written informed consent prior to participation in the trial and who undertake to comply with the protocol.

Exclusion Criteria:

* Patients who are unwilling or unable to be fully evaluated for follow-up.
* Patients who have base AP levels at > 125 IU/L, or levels < 30 IU/L (ammediol, DEA (diethanolamine) units)
* Patients who show pre-operative infections or who are suspected of endocarditis or systemic infection.
* Patients who refuse to accept medically-indicated blood products.
* Patients who have evidence of significant hepatic disease, including history of clinical signs or laboratory values of total bilirubin > 34.2 µmol/L (> 2.0 mg/dL), ALT (>120) or AST (>135) corresponding to > 3X upper limit of normal.
* Patients who received investigational drugs in the 30 days prior to study drug administration, or are currently participating in a study during which the administration of investigational drugs within one month is anticipated.
* Patients who require pre-operative ventilatory support.
* Patients who have renal insufficiency (history of creatinine >177mol/L or >2.0 mg/dL) or chronic renal failure requiring dialysis.
* Patients who are planned to receive leukocyte-depletion filtration as part of the bypass circuitry.
* Patients with severe neurological deficits.
* Patients who have a recent history of drug or alcohol abuse.
* Patients with a diagnosis of idiopathic thrombocytopenia.
* Patients with a history of cancer who have received chemotherapy or radiation therapy within the past 3 months. Patients receiving only adjuvant hormonal therapy are not excluded.
* Patients who are scheduled to receive "stress doses" of glucocorticoids (i.e., doses >2 mg/kg/day of methylprednisolone or equivalent) prior to, during or following surgery.
* Patients who are vegetarians or veganists or those patients that may be expected not to be tolerant for bovine proteins.
* Patients who are, in the opinion of the investigator, unsuitable for the study. A well-documented screening log should be present in the clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
TNF-alpha | one day before till 5 days post surgery
  as indicator of post-surgical inflammatory response

SECONDARY OUTCOMES:
incidence of new organ dysfunctions | till 30 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: M.Erwin S.H. Tan, Prof.Dr.med., Principal Investigator — Catharina Ziekenhuis, Dept. CardioThoracic Surgery
Locations (1):
- Catharina Ziekenhuis, Dept. CardioThoracic Surgery, Eindhoven, Netherlands